CLINICAL TRIAL: NCT00100282
Title: Single Dose Escalation Safety Study of PPI-1019 in Patients With Mild-Moderate Alzheimer's Disease
Brief Title: Safety Study of PPI-1019 in Patients With Mild-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PRAECIS Pharmaceuticals Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1019-03-01
Record Dates: First submitted 2004-12-27; First posted 2004-12-28 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Alzheimer's Disease
Keywords: Mild-moderate Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: PPI-1019 (APAN)

SUMMARY:
This is a multi-center, double-blind, inpatient study followed by outpatient, placebo-controlled, single-dose, dose-escalation evaluation of the safety and tolerability of PPI-1019 in patients with mild-moderate Alzheimer's disease (AD). Up to 12 sequential cohorts of 8 patients (6 active and 2 placebo) will be given a single PPI-1019 dose intravenously (IV) over 1 minute in order to determine a maximum tolerated dose (MTD). The MTD will be the dose immediately below the not-tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Patient has the ability to understand the requirements of the study, provide written informed consent, and abide by the requirements of the study.
* Patient has a caregiver willing to assist the patient's involvement in the study.
* Patient is a male or female between the ages of 50 and 80 with a body mass index (BMI) below 31. Females must be post-menopausal at least

  1 year or surgically sterilized.
* Patient must have a cognitive deficit present for at least one year and meet DSM IV criteria for Alzheimer's Disease and meet National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for the presence of probable Alzheimer's Disease.
* Patient's severity of Alzheimer's disease must be mild-moderate, documented with a Mini Mental State Exam (MMSE) score of 12-26.
* Patient has a computerized tomography (CT) scan or magnetic resonance imaging (MRI) within the prior 12 months which is compatible with a diagnosis of probable AD.
* If a patient is being treated for Alzheimer's disease, it must be with a single agent (donepezil, rivastigmine, galantamine, or memantine) and with a dose which has been stable for at least 3 months.
* Patient is otherwise in good general health. Treatment of hypertension with no more than 2 medications and for hyperlipidemia with one agent is acceptable provided drugs and dosages have been stable for at least 30 days.
* Patient agrees to abstain from alcohol and not take any other drugs, dietary supplements, or herbal therapies other than Mylanta®, ibuprofen, or a multivitamin for the length of the study (screening to follow-up visit Day 22).
* Patient agrees not to donate blood or blood products while participating in this study and for at least 60 days after discontinuing from the study.

Exclusion Criteria:

* Patient has participated in a clinical trial of another investigational drug or device, or has taken any experimental drug within 30 days prior to screening.
* Patient has a history compatible with vascular dementia as evidenced by a score of 5 or greater on the modified Hachinski Ischemia Scale.
* Patient has evidence of clinically significant cardiovascular, renal, hepatic, gastrointestinal, neurological, or metabolic disease within the past 6 months (as determined by medical history, ECG results, chest x-ray, or physical examination). Findings of potential significance must be discussed with an appropriate sponsor clinician (or PRAECIS' designee) prior to patient entry.
* Patient has a systolic blood pressure (sitting) of greater than 150 mmHg, a diastolic (sitting) greater than 95 mmHg, a decrease in systolic blood pressure of more than 30 mmHg upon standing for 2 minutes from a sitting or supine position, or a pulse (sitting or supine) less than 55 or greater than 85.
* Patient has any visual, hearing, or communication disabilities impairing his or her ability to participate in the study.
* Patient intends to use any concomitant medications during the study other than those described in Inclusion Criteria.
* Patient has taken any concomitant medication without the approval of the investigator within 7 days prior to Day 1.
* Patient has tested positive for drugs of abuse (benzodiazepines, narcotics, amphetamines, barbiturates, sedatives, hypnotics, cocaine, phencyclidine, alcohol, or cannabinoids) on drug screening or Day -1.
* Patient has any elevations (> 1.2 x ULN) on screening or Day -1 for ALT, AST, bilirubin, creatinine, blood urea nitrogen, or alkaline phosphatase.
* Patient has any other screening or Day -1 laboratory values outside the normal ranges that are deemed clinically significant by the investigator.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2003-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Clinical (adverse events, vital signs, ECG) and laboratory (chemistry, hematology) parameters
Single dose pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Department of Psychiatry & Human Behavior at the University California, Irvine, Orange, California
  - Global Medical Institutes LLC, Princeton, New Jersey